CLINICAL TRIAL: NCT06721169
Title: Minimally Invasive Treatment of Pilonidal Sinus Disease: Which is Better? Phenol or Laser Ablation
Brief Title: Phenol or Laser: Best Minimally Invasive Treatment for Pilonidal Sinus?
Status: Recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hilmi Bozkurt, Associate Professor, Mersin University
Other Study IDs: 2024/883
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pilonidal Sinus Treatment; Pilonidal Sinus Disorder; Surgical Outcomes
Keywords: Pilonidal Disease, Phenol, Laser Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phenol: Patients with uncomplicated pilonidal sinus disease who receive phenol therapy will be included in this group.
- Lazer ablation: Patients with uncomplicated pilonidal sinus disease who underwent laser ablation will be included in this group.

SUMMARY:
Pilonidal sinus disease is a common condition. There is still ongoing research on the ideal treatment. Pilonidal sinus disease is most common in men between the ages of 20 and 30. For patients with symptoms of pilonidal sinüs (pain, itching and discharge with soiling of underwear) that interfere with their normal daily life, several treatment options have emerged. A hairy body, thick skin, overweight, a deep gluteal cleft, lack of hygiene, sedentarism, repeated chafing and previous familial history are commonly admitted as predisposing factors.

There are various surgical and non-surgical methods for its treatment. Many different surgical techniques have been defined. None of these surgical techniques are defined as 'gold standard'.

For many years, wide excision and secondary healing was the standard approach for pilonidal sinus disease. However, when this method resulted in prolonged healing and restriction of regular activities, various reconstructive methods were developed to demonstrate the disadvantages of secondary healing.

A minimally invasive treatment modality for pilonidal sinüs dissease is excision of the sinus pit(s) followed by application of phenol to the sinus tract. Phenol is a sclerosing agent that destroys the epithelium and debris in the sinus, and is, thus, able to promote healing of the sinus.

Recently, advances in laser technology have made laser ablation of the sinus tract possible. The aim is to destroy and obliterate the sinus tracts with thermal energy produced by the laser probe.

The aim of this prospective observational study was to compare phenolization and laser ablation in the treatment of pilonidal sinus disease.

DETAILED DESCRIPTION:
Pilonidal sinus disease refers to a subcutaneous infection occurring in the gluteal sulcus of the sacrococcygeal region. Although the cause is not clear, it is thought to be related to obesity, hairy body, and deep gluteal sulcus. The incidence of this acquired disease is about 26/100,000 subjects worldwide. The incidence rate among males is 4 times higher than that among females. Pilonidal sinus disease was first de scribed by Herbert Mayo in 1833 as a congenital condition, but is now accepted to be an acquired disease, given its absence in childhood .

Although its cause re mains unknown, the increased hormone levels associated with puberty, the growth of thick hair, long periods of sitting, and friction imparted by tight-fitting clothing may be in play. Other risk factors are hirsutism, obesity, and a family history of the disease. As the cause of the dis ease, hairs falling from head, neck, and back are placed in the intergluteal area and hairs that penetrate the skin initiate foreign body reactions. In the affected area, the hairs are moist, sweaty, and unhygienic, readily trig gering development of the subcutaneous skin cysts and sinuses characteristic of the disease, which (in the gluteal region) present as asymptomatic pits, painful abscesses, or sinuses associated with purulent serous discharge.

The acute phase is characterized by sacral abscess, and during the chronic phase cyst formation or persistent sinus discharge may be observed. At present, no consensus exists regarding the best treatment choice, but conservative treatment can only control the symptoms, and most patients have to undergo operation. Traditional surgery has good success rates; it requires removal of all diseased skin and subcutaneous tissue, including wide excision and healing by secondary intention or reconstructive ("flap") techniques, which results in a long recovery time and a large wound. In recent years, minimally invasive surgical methods for the treatment of SPD (such as endoscopic pilonidal sinus ablation, laser ablation, phenolization, or fibrin glue injection) have improved, reducing wound scarring and pain and shortening the time it takes for patients to return to their normal lives. Surgical success is evaluated by recovery time, the time to return to daily activities, and the complication and recurrence rates.

Patients presenting with pilonidal sinus disease at the Department of General Surgery, Mersin University (Türkiye) were evaluated for participation in this study. Patients aged ≥18 years with symptoms related to pilonidal sinus disease were included in this study. A power analysis was performed using the G*Power (v3.1.7) program to determine the sample size.

Exclusion criteria include the absence of symptoms associated with pilonidal sinus disease, suspicion of an extensive subcutaneous sinus tract network, and the presence of a pilonidal abscess and previous surgery for pilonidal sinus disease, recurrent and complicated pilonidal sinüs disease.

At least 64 patients who meet the inclusion and exclusion criteria will be included in this study. Appropriate surgical procedures will be applied to patients with pilonidal sinus disease who apply to Mersin University Hospital General Surgery Department. The method to be applied will be decided by discussing with the patient.

Data for this study will be collected between November 2024 and November 2025. During this period, data from patients who underwent surgery for pilonidal sinus disease at Mersin University Hospital General Surgery Clinic will be collected. Data will be collected from patients who apply for follow-up on the 1st day, 7th day, 6th month and 12th month after laser ablation or phenol treatment. Demographic characteristics, symptoms, clinical examination findings, surgical findings, postoperative VAS pain scores, wound complications, recurrence rates and return to daily life times will be examined. This data will be obtained through the retrospective review of medical records and confirmed by face-to-face interviews with patients who have attended the outpatient clinic, and then recorded in the data collection form.

Data collection will continue until at least 32 patients are reached in the phenolization and laser ablation groups. Once the target sample size is reached, new data collection from patients will be terminated and statistical analyses will be performed to compare prevalence between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older with pilonidal sinus disease
* Patients who have not had any previous treatment for pilonidal sinus disease
* Patients with uncomplicated pilonidal sinus
* Having been diagnosed with pilonidal sinus disease
* Patients whose descriptive and clinical characteristics are recorded in their medical files
* Those who have signed the Informed Voluntary Consent Form/Written Consent Form

Exclusion Criteria:

* Patients who have previously been treated for pilonidal sinus disease
* Patients with complicated pilonidal sinus disease
* Patients aged under 18
* Patients whose descriptive and clinical characteristics are not recorded in their file records
* Those who have not signed the Informed Voluntary Consent Form/Written Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will be conducted at the Department of General Surgery, Mersin University Hospital between December 15, 2024 and December 15, 2025. The study population consists of adult patients (≥18 years old) diagnosed with pilonidal sinus disease who are scheduled for surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 7 day
  Postoperative complications will be assessed during a 7-day follow-up period. All complications will be documented during hospitalization and at scheduled follow-up visits, including surgical site infections, bleeding, and pulmonary complications.

SECONDARY OUTCOMES:
Length of Hospital Stay | 7 day
  The duration of hospitalization will be measured from the day of surgery until discharge, with standardized discharge criteria including adequate pain control, successful oral intake and return of bowel function
Return to Daily Activities | 7 day
  The evaluation of the patients' return to their initial functional status will be evaluated using standardized questionnaires, either in person during outpatient clinic visits or over the phone (in cases where they do not come for regular follow-ups). This involves monitoring the time required to resume basic activities of daily living (ADLs) and reach preoperative functional capacity.
Recurrence of disease | 1 year
  Patients will be evaluated using standard questionnaires during their 6-month and 1-year outpatient clinic visits or by phone (in cases where they do not come for regular follow-ups). Patients will be evaluated for symptoms of recurrence (discharge, pain, abscess, new pit formation).

CONTACTS AND LOCATIONS:
Overall Officials: Doğuş Parlak, PhD, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data underlying the primary and secondary outcomes of the study, including demographics (age, gender, BMI), clinical parameters (pain, discharge, infection), surgical details, and postoperative outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be accessible from 6 months to 36 months after the publication of the article. Data access will be granted to researchers who submit a methodologically sound proposal and receive approval from an independent review committee. Proposals should be directed to the Mersin University Hospital Department of General Surgery.
Access Criteria: To gain access, researchers will be required to sign a data access agreement and, if necessary, obtain relevant ethics approval. The study protocol, statistical analysis plan, informed consent form and clinical study report will also be provided. Data will be shared via a secure online platform with appropriate confidentiality and security measures in place.

REFERENCES:
- [Background] Romic I, Augustin G, Bogdanic B, Bruketa T, Moric T. Laser treatment of pilonidal disease: a systematic review. Lasers Med Sci. 2022 Mar;37(2):723-732. doi: 10.1007/s10103-021-03379-x. Epub 2021 Jul 22. PMID 34291332
- [Background] Yardimci VH. Outcomes of Two Treatments for Uncomplicated Pilonidal Sinus Disease: Karydakis Flap Procedure and Sinus Tract Ablation Procedure Using a 1,470 nm Diode Laser Combined With Pit Excision. Lasers Surg Med. 2020 Nov;52(9):848-854. doi: 10.1002/lsm.23224. Epub 2020 Feb 17. PMID 32064640
- [Background] Elvira Lopez J, Escuder Perez J, Sales Mallafre R, Feliu Villaro F, Caro Tarrago A, Espina Perez B, Ferreres Serafini J, Jorba Martin R. Randomised clinical trial to test the phenolization in sacrococcygeal pilonidal disease. Int Wound J. 2023 Aug;20(6):2181-2189. doi: 10.1111/iwj.14096. Epub 2023 Jan 26. PMID 36700412
- [Background] Pronk AA, Smakman N, Furnee EJB. Short-term outcomes of radical excision vs. phenolisation of the sinus tract in primary sacrococcygeal pilonidal sinus disease: a randomized-controlled trial. Tech Coloproctol. 2019 Jul;23(7):665-673. doi: 10.1007/s10151-019-02030-w. Epub 2019 Jul 5. PMID 31278458
- [Background] Li Z, Jin L, Gong T, Qin K, Cui C, Wang Z, Wu J. An effective and considerable treatment of pilonidal sinus disease by laser ablation. Lasers Med Sci. 2023 Mar 1;38(1):82. doi: 10.1007/s10103-023-03741-1. PMID 36856904